CLINICAL TRIAL: NCT00801502
Title: The Effects of Oily Fish in Pregnancy on Markers and Manifestations of Allergic Diseases in Infants at Risk of Atopy
Brief Title: Salmon in Pregnancy Study
Acronym: SiPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RHMNUT0044
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Dermatitis; Allergies; Asthma
Keywords: Omega-3; Oily fish; Antioxidant; Selenium; Atopic disease; Pregnancy; Nutrient status
MeSH Terms: conditions — Dermatitis; Hypersensitivity; Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): No change in diet
  Interventions: Other: Control
- Oily fish (Active Comparator): Two portions of salmon per week from week 20 of pregnancy until giving birth
  Interventions: Dietary Supplement: Oily fish consumption

INTERVENTIONS:
Dietary Supplement: Oily fish consumption — Two portions of salmon per week from week 20 of pregnancy until giving birth
  Arms: Oily fish
Other: Control — No change to habitual diet from week 20 of pregnancy until giving birth
  Arms: Control

SUMMARY:
The number of infants and children with allergic disease (dermatitis, allergies, asthma) has increased over the last several decades. This may be related to changes in diet. It is now thought that children become sensitised to allergens very early in life maybe even before they are born. Some studies show that a high omega-3 fat intake by mothers decreases risk of sensitisation in their babies. There is a biological mechanism to explain this. Omega-3 fats are found in oily fish like salmon. In the UK pregnant women are recommended to eat oily fish twice per week. However, consumption of oily fish is known to be low in pregnant women in the UK. This study sets out to identify the effects of increasing salmon intake in pregnant women. The hypothesis being investigated is that : increased consumption of oily fish during pregnancy by women at risk of having offspring who will develop atopy will increase their omega-3 fat and antioxidant status and that of their developing baby and will ameliorate the development of atopic markers and manifestations in the infants.

DETAILED DESCRIPTION:
The prevalence of childhood atopic diseases (eczema, rhinitis [hay-fever], asthma, allergies) has increased dramatically over the last 30 years or so. This must be due to environmental changes. Dietary change is believed to be an important causative factor and three diet related hypotheses have been proposed. The first of these ("the PUFA hypothesis") is that the increase in intake of n-6 polyunsaturated fatty acids (PUFA) over the last 30 years has resulted in an absolute and relative decline in intake of n-3 PUFA, especially long chain n-3 PUFA. There is a plausible biological mechanism whereby a high n-6 to n-3 PUFA ratio would skew the immune system to favour sensitisation to allergens. The second diet hypothesis ("the antioxidant hypothesis") is that there is a lower status of antioxidant vitamins and minerals than 30 years ago and that the resulting increased oxidant stress skews the immune system to favour sensitisation to allergens. The third diet hypothesis ("the gut microflora hypothesis") is that the maturing microflora within the intestinal tract of the neonate plays a role in development of atopy through interactions with the gut immune system. Factors that influence development of neonatal gut microflora include maternal gut microflora and infant diet (e.g. breast milk composition). Since maternal diet will affect maternal gut microflora and also breast milk composition a link is suggested between modification of the maternal diet in pregnancy and development of atopy in the infant through an effect on gut microflora.

It is now recognised that sensitisation to the allergens that trigger atopic disease occurs early in life, and in many cases in utero [4]. Thus, it is most likely maternal diet during pregnancy that is important in influencing risk of atopic disease in children. There is much evidence that n-3 PUFA status is lower in plasma, erythrocytes, white cells and milk of mothers of atopic children and also in umbilical cord plasma and erythrocytes [5]. Likewise, the status of some antioxidant minerals (e.g. Se) in cord blood has been reported to be lower in children who went on to develop atopic disease than in those who did not. Finally, atopic infants have a different gut microflora than non-atopic infants. These studies suggest that maternal status of n-3 PUFA and antioxidants, and possible of certain gut microbes, is important in determining atopic outcome in children. Not surprisingly therefore, there is substantial interest in supplementation studies in pregnant women, particularly those whose babies are at risk of atopic disease (e.g. from a family history). Fish, especially oily fish like salmon, and fish oil are very good sources of long chain n-3 PUFA. A recent study investigating the effect of fish oil supplementation in pregnant women reported an alteration in the cytokine profile of umbilical cord plasma that is consistent with protection towards atopy. The study went on to demonstrate a reduced severity of atopic dermatitis and a decreased likelihood of skin-prick positivity to a variety of common allergens in the children at one year of age. Oily fish represent a unique opportunity to reduce atopy risk because they are rich sources of both n-3 PUFA and antioxidant minerals (Se). They represent a more attractive option than supplementation with fish oil capsules. Pregnant women have a low intake of fish. Current UK recommendations are that "women of reproductive age should aim to consume within the range of one to two portions of oily fish a week". The upper limit of this range is below that for the recommendations made for boys, men and women not of reproductive age. This is because of concern about contaminants in some species of oily fish (e.g. tuna). Aquaculture producing salmon with low contaminant levels is therefore an ideal solution to enable oily fish consumption by pregnant women. Consumption of tailor-made salmon by pregnant women could prevent the development of atopic disease in their children. It is important that this be assessed through a well-designed and rigorous intervention study relating maternal oily fish consumption to atopic disease in the offspring, at the same time assessing effects of maternal fish consumption on fetal growth and maternal and fetal body composition.

Hypothesis:

Increased consumption of oily fish during pregnancy by women at risk of having offspring who will develop atopy will increase their n-3 PUFA and antioxidant status and that of their developing baby and will ameliorate the development of atopic markers and manifestations in the infants.

Objectives:

1. To conduct a dietary intervention study in pregnant women using long chain n-3 PUFA-rich salmon.
2. To determine the effects of increased consumption of oily fish during pregnancy on fetal growth and adaptations and on maternal and fetal body composition.
3. To determine the effects of increased consumption of oily fish during pregnancy on maternal and fetal (i.e. cord blood) nutrient status
4. To determine the effects of increased consumption of oily fish during pregnancy on maternal and fetal (i.e. cord blood) immune status
5. To determine the effects of increased consumption of oily fish during pregnancy on predictors of atopic disease in cord blood, and on the development of atopic disease in infancy.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women before 19 weeks gestation, with healthy uncomplicated singleton pregnancies, but whose babies are at risk of atopy (i.e. one or more first degree relatives affected).
2. Not habitual consumers of oily fish (< 2 portions of oily fish per month excluding tinned tuna).
3. Not using fish oil supplements (currently or in the last 3 months)
4. Age 18-40 y.

Exclusion Criteria:

1. Habitual consumer of oily fish (> 2 portions of oily fish per month excluding tinned tuna).
2. Use of fish oil supplements within the previous 3 months.
3. Not willing for essential identifiable information being stored for tracking purposes.
4. Participation in another research study.
5. Known diabetic and/or other auto-immune disease, e.g. SLE, MS, Thyroid Disease.
6. Adults with learning disabilities.
7. Adults who have a terminal illness.
8. Adults with mental health problems.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Omega-3 fatty acid status in maternal and umbilical cord plasma | Weeks 20, 34 and 38 of pregnancy and at birth (in cord)

SECONDARY OUTCOMES:
Antioxidant status in maternal and umbilical cord blood | Weeks 20, 34 and 38 of pregnancy and at birth (in cord)
Allergic sensitisation of infants | 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Calder, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom

REFERENCES:
- [Background] Garcia-Rodriguez CE, Helmersson-Karlqvist J, Mesa MD, Miles EA, Noakes PS, Vlachava M, Kremmyda LS, Diaper ND, Godfrey KM, Calder PC, Gil A, Basu S. Does increased intake of salmon increase markers of oxidative stress in pregnant women? The salmon in pregnancy study. Antioxid Redox Signal. 2011 Dec 1;15(11):2819-23. doi: 10.1089/ars.2011.4108. Epub 2011 Jul 22. PMID 21689025
- [Background] Miles EA, Noakes PS, Kremmyda LS, Vlachava M, Diaper ND, Rosenlund G, Urwin H, Yaqoob P, Rossary A, Farges MC, Vasson MP, Liaset B, Froyland L, Helmersson J, Basu S, Garcia E, Olza J, Mesa MD, Aguilera CM, Gil A, Robinson SM, Inskip HM, Godfrey KM, Calder PC. The Salmon in Pregnancy Study: study design, subject characteristics, maternal fish and marine n-3 fatty acid intake, and marine n-3 fatty acid status in maternal and umbilical cord blood. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1986S-1992S. doi: 10.3945/ajcn.110.001636. Epub 2011 Aug 17. PMID 21849598
- [Background] van den Elsen LW, Noakes PS, van der Maarel MA, Kremmyda LS, Vlachava M, Diaper ND, Miles EA, Eussen SR, Garssen J, Willemsen LE, Wilson SJ, Godfrey KM, Calder PC. Salmon consumption by pregnant women reduces ex vivo umbilical cord endothelial cell activation. Am J Clin Nutr. 2011 Dec;94(6):1418-25. doi: 10.3945/ajcn.111.016592. Epub 2011 Oct 19. PMID 22011457
- [Background] Helmersson-Karlqvist J, Miles EA, Vlachava M, Kremmyda LS, Noakes PS, Diaper ND, Godfrey KM, Calder PC, Basu S. Enhanced prostaglandin F2alpha formation in human pregnancy and the effect of increased oily fish intake: results from the Salmon in Pregnancy Study. Prostaglandins Leukot Essent Fatty Acids. 2012 Jan-Feb;86(1-2):35-8. doi: 10.1016/j.plefa.2011.10.008. Epub 2011 Nov 1. PMID 22047909
- [Background] Noakes PS, Vlachava M, Kremmyda LS, Diaper ND, Miles EA, Erlewyn-Lajeunesse M, Williams AP, Godfrey KM, Calder PC. Increased intake of oily fish in pregnancy: effects on neonatal immune responses and on clinical outcomes in infants at 6 mo. Am J Clin Nutr. 2012 Feb;95(2):395-404. doi: 10.3945/ajcn.111.022954. Epub 2012 Jan 4. PMID 22218160
- [Background] Garcia-Rodriguez CE, Mesa MD, Olza J, Vlachava M, Kremmyda LS, Diaper ND, Noakes PS, Miles EA, Ramirez-Tortosa MC, Liaset B, Froyland L, Rossary A, Farges MC, Vasson MP, Aguilera CM, Helmersson-Karlqvist J, Godfrey KM, Calder PC, Basu S, Gil A. Does consumption of two portions of salmon per week enhance the antioxidant defense system in pregnant women? Antioxid Redox Signal. 2012 Jun 15;16(12):1401-6. doi: 10.1089/ars.2012.4508. Epub 2012 Feb 21. PMID 22229304
- [Background] Garcia-Rodriguez CE, Olza J, Aguilera CM, Mesa MD, Miles EA, Noakes PS, Vlachava M, Kremmyda LS, Diaper ND, Godfrey KM, Calder PC, Gil A. Plasma inflammatory and vascular homeostasis biomarkers increase during human pregnancy but are not affected by oily fish intake. J Nutr. 2012 Jul;142(7):1191-6. doi: 10.3945/jn.112.158139. Epub 2012 May 23. PMID 22623389
- [Background] Urwin HJ, Miles EA, Noakes PS, Kremmyda LS, Vlachava M, Diaper ND, Perez-Cano FJ, Godfrey KM, Calder PC, Yaqoob P. Salmon consumption during pregnancy alters fatty acid composition and secretory IgA concentration in human breast milk. J Nutr. 2012 Aug;142(8):1603-10. doi: 10.3945/jn.112.160804. Epub 2012 Jun 27. PMID 22739373
- [Background] Urwin HJ, Miles EA, Noakes PS, Kremmyda LS, Vlachava M, Diaper ND, Godfrey KM, Calder PC, Vulevic J, Yaqoob P. Effect of salmon consumption during pregnancy on maternal and infant faecal microbiota, secretory IgA and calprotectin. Br J Nutr. 2014 Mar 14;111(5):773-84. doi: 10.1017/S0007114513003097. Epub 2013 Oct 16. PMID 24128654
- [Background] Rossary A, Farges MC, Lamas B, Miles EA, Noakes PS, Kremmyda LS, Vlachava M, Diaper ND, Robinson SM, Godfrey KM, Calder PC, Vasson MP. Increased consumption of salmon during pregnancy partly prevents the decline of some plasma essential amino acid concentrations in pregnant women. Clin Nutr. 2014 Apr;33(2):267-73. doi: 10.1016/j.clnu.2013.04.013. Epub 2013 May 1. PMID 23684555